CLINICAL TRIAL: NCT04793867
Title: Regional Phenotyping of Cystic Fibrosis Lung Disease and Non-CF Bronchiectasis
Brief Title: Regional Phenotyping of CF and Non-CF Bronchiectasis
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Zackary I. Cleveland, PhD, Principal Investigator, Children's Hospital Medical Center, Cincinnati
Other Study IDs: 2020-0814
Record Dates: First submitted 2021-02-23; First posted 2021-03-11 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cystic Fibrosis; Non-CF Bronchiectasis
Keywords: Cystic Fibrosis; hyperpolarized xenon; LCI; Non-CF Bronchiectasis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Xenon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CF and Non-CF Bronchiectasis: In the first arm (Aims 1 & 2) Up to 50 subjects will be recruited-approximately 25 with normal FEV1 (>85% predicted) and 25 with mild to moderate disease. All subjects will be asked to undergo longitudinal (i.e., approximately annually) 129Xe and UTE MRI, spirometry, and lung clearance index (LCI) measurement.
  Interventions: Drug: Xenon
- Healthy Subjects: Up to 50 age and sex matched control subjects (i.e., subjects with no known cardiopulmonary disorders) may also be recruited to provide a reference data set from healthy subjects for comparison.
  Interventions: Drug: Xenon

INTERVENTIONS:
Drug: Xenon — Subjects will be scanned on a commercial 3T whole-body MRI scanner equipped with high-performance gradient systems. Natural isotopic abundance or isotopically-enriched xenon gas (~86% 129Xe, Linde Inc.) will be used for all studies. Subjects will be positioned supine in the scanner with a 129Xe RF coil around their chests. Using conventional proton MRI and a breath-hold acquisition, "scout" images will be obtained to localize the subject for subsequent 129Xe acquisitions. 129Xe images will be acquired using the same breath-hold maneuver and a pulse sequence, covering the entire lung (acquisition time <10 s, approximately 3-mm in-plane resolution, 15-mm slice thickness or less). Additional scans (sequences) may be performed. A maximum of 4 doses of 129Xe will be given throughout the study following the calibration dose.
  Other Names: 129Xe

SUMMARY:
The Investigators propose to study pediatric subjects who are diagnosed with cystic fibrosis (CF) and patients with non-CF bronchiectasis, with the goal of developing markers of CF lung disease severity, progression, and therapy response. The Investigator's central hypothesis is that image-based markers can forecast pathophysiology prior to spirometric changes.

DETAILED DESCRIPTION:
Specific Aim 1: Validate functional imaging markers in CF patients with normal spirometry but abnormal ventilation. The Investigators hypothesize imaging phenotype can predict lung function decline, even in CF patients with normal spirometry. The Investigators will test this hypothesis by performing annual HP 129Xe ventilation MRI in a cohort of CF patients of which a subset has normal FEV1 (≥85% predicted) at baseline.

Specific Aim 2: Determine the sensitivity and specificity of early structural remodeling in CF lung disease. The Investigator's preliminary studies show that imaging markers of structural lung remodeling can be measured via radiation-free MRI (as opposed to x-ray CT). We assess the sensitivity to identify subjects with irreversible remodeling by performing serial ultra-short UTE MRI.

In the first arm (Aims 1 & 2) Up to 50 subjects will be recruited-approximately 25 with normal FEV1 (>85% predicted) and 25 with mild to moderate disease. All subjects will be asked to undergo longitudinal (i.e., approximately annually) 129Xe and UTE MRI, spirometry, and lung clearance index (LCI) measurement. If possible, studies will be coordinated with clinical visits to maximize recruitment and retention. Up to 50 age and sex matched control subjects (i.e., subjects with no known cardiopulmonary disorders) may also be recruited to provide a reference data set from healthy subjects for comparison.

Healthy adults, including CCHMC employees) and children >5 years old may be recruited as needed for MRI sequence development and validation.

In the second arm (Aim 3), 50 CF patients with bronchiectasis and 50 with non-CF bronchiectasis will be recruited from patients already undergoing clinical bronchoscopies. Before bronchoscopy, subjects will undergo UTE. BAL will be obtained from radiologically normal areas and regions with abnormalities. (Note, image-guided sampling from multiple sites is routine practice at CCHMC in patients with CF and non-CF bronchiectasis. As such, the proposed studies will not alter the sampling pattern in a clinically significant way or increase procedure time, and will thus add no patient risk.) Clinical BAL will be collected from these regions, and small aliquots (~500 µL) will be stored separately for proteomics. The remaining fluid will be pooled and submitted for routine clinical testing, with ~500 µL reserved for pooled proteomics. The Investigators will recruit ~10 subjects/yr from both CF and non-CF groups, who will be followed annually with UTE and proteomic analysis that will be collected under Dr. Ziady's companion protocol, titled Proteomic biomarkers of CF disease and non-CF bronchiectasis to measure prognostic markers of disease-in particular of persistent bronchiectasis. For all subjects, clinical data (e.g., age, gender, CF genotype, microbiology, therapies-including CFTR modulators-and exacerbation frequency) will be captured in a REDcap database.

ELIGIBILITY:
Inclusion Criteria:

* CF Patients: Diagnosis of CF based on sweat chloride >60 mMol/l
* Presence of two disease causing CFTR mutations, or end organ manifestations of disease.
* Age minimum 5 years.
* Care provided by the CCHMC CF Care Center or other regional CF Care Centers if required to achieve recruitment goals.

Exclusion Criteria:

* Patients meeting standard MRI exclusions criteria (non-MRI-compatible metal implants, claustrophobia, etc.)
* Pregnancy or lactation.

Inclusion Criteria of Healthy Subjects:

* Subjects 5 years of age and older with no known history of cardiopulmonary disease.

Exclusion Criteria of Healthy Subjects:

* Patients meeting standard MRI exclusions criteria (non-MRI-compatible metal implants, claustrophobia, etc.)
* Pregnancy or lactation.

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: CF and Non-CF Bronchiectasis patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of ventilated volume predictions obtained with 129Xe MRI vs 1H MRI | Annually for 5 years
  Quantify the measurement agreement between the ventilated volume of CF and Non-CF Bronchiectasis lungs vs healthy lungs

CONTACTS AND LOCATIONS:
Overall Officials: Zackary I Cleveland, PhD, Principal Investigator — CCHMC
Locations (1):
- Penny New, Cincinnati, Ohio, United States